CLINICAL TRIAL: NCT00230958
Title: Randomized, Double-Blind, Multicenter Study to Compare the Safety and Efficacy of Viramidine to Ribavirin in Treatment-Naive Patients With Chronic Hepatitis C
Brief Title: Study of Viramidine to Ribavirin in Patients With Chronic Hepatitis C Who Are Treatment-Naive
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RNA003142-301
Record Dates: First submitted 2005-09-29; First posted 2005-10-03 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Chronic Hepatitis C
Keywords: Viramidine; Ribavirin; Valeant; Hepatitis C; Pegylated interferon alfa-2b
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — taribavirin; Ribavirin; peginterferon alfa-2b

INTERVENTIONS:
Drug: Viramidine
Drug: Ribavirin
Drug: pegylated interferon alfa-2b

SUMMARY:
This purpose of this study is to determine the safety and effectiveness of viramidine to ribavirin in chronic hepatitis C patients who have never before recieved treatment.

DETAILED DESCRIPTION:
Compare the efficacy and safety of viramidine 600 mg BID versus ribavirin 1000/1200 mg/day, both drugs administered in combination with pegylated interferon alfa-2b to treatment-naive patients with chronic hepatitis C (CHC)

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naive patients with compensated chronic hepatitis C.
* HCV RNA >2000 copies/mL (780 IU/mL) as determined by NGI SuperQuant serum HCV RNA quantification, with a lower limit of detection of 100 copies/mL (39 IU/mL).

Exclusion Criteria:

* Severe neuropsychiatric disorders
* History or clinical manifestations of significant metabolic, hematological, pulmonary, ischemic heart disease, significant or unstable heart disease, gastrointestinal, neurological, renal, urological, endocrine, opthalmologic disorders including severe retinopathy, or immune mediated disease
* Pregnant or breast-feeding patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900
Dates: Start 2003-12; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
- Efficacy: Undetectable plasma HCV RNA (less than 100 copies/mL) at the end of the 24-week post-treatment follow-up period.
- Safety: The proportion of patients with hemoglobin less than 10 g/dL at any time during treatment or at least 2.5 g/dL drop from baseline.

SECONDARY OUTCOMES:
- Efficacy: Undetectable plasma HCV RNA at treatment week 24
- Efficacy: Undetectable or at least a 2-log drop from baseline at treatment weeks 12 and 24
- Safety: Monitoring of adverse events
- Safety: Monitoring of abnormal changes in laboratory parameters that are not disease-related

CONTACTS AND LOCATIONS:
Overall Officials: Ralph T. Doyle, Study Director — Bausch Health Americas, Inc.